CLINICAL TRIAL: NCT00902356
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 167 in Healthy Men and Postmenopausal Women
Brief Title: A First-in-human Study Evaluating AMG 167 in Healthy Men and Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080049
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Osteopenia
Keywords: Amgen; Phase 1; First in Human; Postmenopausal
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- B (Active Comparator): Six female subjects in each of cohorts 1 to 5 will receive AMG 167; six male subjects in each of cohorts 6 and 8; three female subjects in each of cohorts 7 and 9.
  Interventions: Drug: Placebo
- A (Placebo Comparator): Two female subjects in each of cohorts 1 to 5 will receive placebo; two male subjects in each of cohorts 6 and 8; and 1 female subject in each of cohorts 7 and 9.
  Interventions: Drug: AMG 167

INTERVENTIONS:
Drug: AMG 167 — Subjects will be randomized to receive 1 of 5 doses of AMG 167 or equivalent volume of placebo administered as a single dose. Postmenopausal women will receive AMG 167 in fixed doses of 21 mg, 70, 210, 350, or 700 mg SC (under the skin), or 70 mg or 350 mg IV (in the vein), while men will receive doses of 70 mg or 350 mg SC or IV.
  Arms: A
Drug: Placebo — Subjects will be randomized to receive 1 of 5 doses of AMG 167 or equivalent volume of placebo administered as a single dose. Postmenopausal women will receive AMG 167 in fixed doses of 21 mg, 70, 210, 350, or 700 mg SC (under the skin), or 70 mg or 350 mg IV (in the vein), while men will receive doses of 70 mg or 350 mg SC or IV.
  Arms: B

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of AMG 167 following a single dose subcutaneous (SC) or intravenous (IV) administration in healthy men and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 45 to 65 years of age
* Postmenopausal females defined as 12 continuous months of spontaneous amenorrhea confirmed by a serum follicle-stimulating hormone (FSH) result > 40mIU/mL, or at least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy)
* Men must agree to use highly effective methods of contraception; males must agree to not donate sperm for the entire study and 7 months after the end of treatment
* Weight ≤ 98 kg (216 lb) and/or height ≤ 196 cm (77 in)
* Has no history or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Negative urine screen for potential drugs of abuse at screening and admission, unless medication is prescribed by a physician

Exclusion Criteria:

* Healthy males with partners who are pregnant at the time of screening; or healthy males with partners who plan to become pregnant during the study
* Osteoporosis, as defined by BMD t-scores of the lumbar spine (L1-L4) or total evaluable vertebrae; or femoral neck ≤ 2.5
* Diagnosed with any condition that will affect bone metabolism
* Diagnosis of clotting factor deficiency or history of bleeding or coagulation disorder (including history of heparin or warfarin administration)
* Subjects with fewer than 2 evaluable vertebrae; metal in hips bilaterally that would not allow for at least one evaluable hip; metal in forearms bilaterally that would not allow for at least one evaluable forearm
* Abnormal international normalized ratio or partial thromboplastin time
* Administration of the following medications within 6 months before study drug administration:
* Hormone replacement therapy [Infrequent use of estrogen vaginal creams (< 3 times per week) is allowed.]
* Calcitonin
* Parathyroid hormone (or any derivative)
* Supplemental Vitamin D > 1,000 IU/day
* Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed)
* Anabolic steroids
* Calcitriol, and available analogues
* Administration of the following medications within 12 months before study drug administration:
* Bisphosphonates
* Fluoride for osteoporosis
* Administration of herbal medications within 2 weeks or 5 half-lives (whichever is longer) before study drug administration
* Greatly differing levels of physical activity or constant levels of intense physical exercise during the 6 months before study drug administration
* Known alcohol abuse or use of illicit drugs within 12 months of admission
* Unwilling or unable to limit alcohol consumption throughout the course of the study
* Known sensitivity to mammalian-derived drug preparations
* Known to be hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus positive, or a known diagnosis of acquired immunodeficiency syndrome
* An unstable medical condition, defined as having been hospitalized within 28 days before day -1, major surgery within 6 months before day -1, or otherwise unstable in the judgment of the investigator
* Has any clinically significant abnormality during the screening physical examination, ECG, or laboratory evaluation
* Unavailable for follow-up assessment or any concerns for subject's compliance with the protocol procedures
* Any other condition that might reduce the chance of obtaining data required by the protocol or that might compromise the ability to give truly informed consent
* Has participated in another clinical study within 4 weeks of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known
* Has donated or lost 400 mL or more of blood or plasma within 8 weeks of study drug administration
* Previous exposure to AMG 785

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The number (percent) of subjects reporting treatment-emergent adverse events. | Cohort 1 - 29 days; cohorts 2, 3, 6, and 7 - 57 days; cohorts 4, 5, 8, and 9 - 85 days
The number of subjects experiencing clinically significant changes in safety laboratory tests, physical examinations, vital signs, or electrocardiograms (ECGs). | Cohort 1 - 29 days; cohorts 2, 3, 6, and 7 - 57 days; cohorts 4, 5, 8, and 9 - 85 days
The number of subjects who develop anti-AMG 167 antibodies. | Cohort 1 - 29 days; cohorts 2, 3, 6, and 7 - 57 days; cohorts 4, 5, 8, and 9 - 85 days

SECONDARY OUTCOMES:
Pharmacokinetic and phamacodynamic parameters [serum procollagen type 1 N-terminal propeptide (P1NP), BSAP, osteocalcin, sCTX, sclerostin levels, and bone mineral density (BMD) for higher dose levels] after single dose SC or IV administration of AMG 167. | Cohort 1 - 29 days; cohorts 2, 3, 6, and 7 - 57 days; cohorts 4, 5, 8, and 9 - 85 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com